CLINICAL TRIAL: NCT01754285
Title: A Randomized, Double-Blind, Double Dummy, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy of LF-PB 10 mg, 20 mg, and 30 mg to Treat Lymphorrhea Post Axillary Dissection in Breast Cancer
Brief Title: Extended-release of Octreotide (LF-PB) for the Treatment of Lymphorrhea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chemi S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LF-PB/11/04
Record Dates: First submitted 2012-12-12; First posted 2012-12-21 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Lymphorrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- LF-PB 10 mg (Experimental): 2 IM injections = placebo + 10 mg
  Interventions: Drug: LF-PB and Placebo
- LF-PB 20 mg (Experimental): 2 IM injections = placebo + 20 mg
  Interventions: Drug: LF-PB and Placebo
- LF-PB 30 mg (Experimental): 2 IM injections = 10 mg + 20 mg
  Interventions: Drug: LF-PB
- Placebo (Placebo Comparator): 2 IM injections of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LF-PB and Placebo
  Other Names: extended-release of octreotide and placebo
  Arms: LF-PB 10 mg; LF-PB 20 mg
Drug: Placebo
  Arms: Placebo
Drug: LF-PB
  Other Names: LF-PB 10 mg and LF-PB 20 mg
  Arms: LF-PB 30 mg

SUMMARY:
This is a phase II, multicenter, double-blind, double-dummy, parallel-group, placebo-controlled, study to evaluate LF-PB versus placebo in female patients with brest cancer who are undergoing breast surgery with axillary lymphnode dissection.

Recruited patients will be randomly assigned to one of the following treatment groups: Placebo, LF-PB 10 mg, LF-PB 20 mg and LF-PB 30 mg.

Mode of administration is single intramuscular (IM) injection so the treatments arms are as follows:

Placebo: 2 injections of placebo LF-PB 10 mg: 2 injections = placebo + 10 mg LF-PB 20 mg: 2 injections = placebo + 20 mg LF-PB 30 mg: 2 injections = 10 mg + 20 mg

The study will randomize a total of 120 patients (30 per arm) in about 10 Italian Sites.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged 18 to 80 years inclusive
2. Body mass index (BMI) ≥18 kg/m2
3. Signed informed consent form
4. Diagnosis of BC
5. Undergoing breast surgery with ALND Note: Collagen powder or fibrin sealant are not permitted.
6. Negative serum pregnancy test for women of childbearing potential Note: Female patients of child-bearing potential should be advised to use adequate contraception if necessary during treatment with octreotide.
7. AST and alanine aminotransferase ALT <1.5 x the upper limit of normal
8. Ability to fully understand all study procedures and to comply with study visits scheduled for the duration of the study.

Exclusion Criteria:

1. Presence of any of the following conditions:

   1. Previous axillary surgery on the same armpit undergoing surgery in this study
   2. Previous chemotherapy or radiotherapy within five years from study drug administration
   3. Previous neoadjuvant therapy
   4. Recurrent BC on the same breast undergoing surgery in this study
   5. Diabetes
   6. Cholelithiasis
   7. Hypothyroidism. If patient is being administered Euritox/ Levothyroxine (or analogues) and levels of T3, T4 and TSH are confirmed to be within the normal ranges at screening, the patient can be enrolled in this study.
   8. Hepatitis
   9. Pregnant or lactating
   10. Human immunodeficiency virus or hepatitis B or C by screening serology
2. History of radiotherapy on the same breast or armpit undergoing surgery in this study.
3. History of anaphylaxis to study drug
4. Ascertained or presumptive hypersensitivity to the active principle and/or the ingredients of the study drug formulation
5. QTc interval extension at screening or baseline > 450 msec (as the mean of 3 consecutive readings 5 minutes apart)
6. Presence of any disease or use of concomitant medication known to increase the QT interval (see Appendix 2 for a list of such compounds)
7. Clinically significant or relevant abnormal medical history, vital sign, physical examination, ECG, or laboratory evaluation finding
8. Current or recurrent disease that could affect the results of the clinical or laboratory assessments required for the study

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2012-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
effect of LF-PB 10 mg, 20 mg, and 30 mg on time to resolution of lymphorrhea; | 12 weeks post surgery
  End of lymphorrhea will be declared when the lymph volume measured by the patient is < 50 ml/day in 2 consecutive days.
number of AEs and laboratory, ECG, vital sign abnormalities of LF-PB 10 mg, 20 mg, and 30 mg | 12 weeks after surgery
  Safety and tolerability of LF-PB

SECONDARY OUTCOMES:
effects of LF-PB 10, 20, and 30 mg on the daily volume of lymph collected from the drain | 12 weeks after surgery
  daily volume of lymph collected from the drain
number of complications related to lymphorrhea | 12 weeks after surgery
  effect of LF-PB 10, 20 and 30 mg on complications related to lymphorrhea
PK profile (Cmax, Tmax, AUC0-t and possibly AUC0-inf and T1/2) of LF-PB 10, 20 and 30 mg | 12 weeks after surgery
  PK parameters

OTHER OUTCOMES:
correlation between LF-PB exposures and efficacy after the administration of LF-PB 10 mg, 20 mg, and 30 mg | 12 weeks after surgery
  correlation between exposure of the drug and efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Carcoforo, MD, Principal Investigator — Clinica Chirurgica, Azienda Ospedaliero-Universitaria Arcispedale "S. Anna" Ferrara
Locations (13):
- Italy (13):
  - Humanitas Centro Catanese di Oncologia Dipartimento di Oncologia -Chirurgia Oncologica Generale, Via V.E. Dabormida, 64, Catania
  - Fondazione per la Ricerca e la Cura dei Tumori "Tommaso Campanella" Unità Operativa Complessa CRR per il Counselling Genetico e le Terapie Innovative in Oncologia Medica, Viale Europa-Loc. Germaneto, Catanzaro
  - Azienda Ospedaliera OIRM Sant'Anna Dipartimento Funzionale di Oncologia - Breast Unit, Corso Spezia, 60 Torino
  - IRCCS Azienda Ospedaliero Universitaria San Martino di Genova - IST Genova Dipartimento Chirurgia Ospedaliera - Semeiotica Chirurgica e Chirurgia Senologica, L.go Rosanna Benzi,10 Genova
  - Azienda Ospedaliero Universitaria Consorziale Policlinico di Bari Chirurgia Generale Universitaria "G.Marinaccio", Piazza Giulio Cesare 11 Bari
  - Azienda Ospedaliero-Universitaria Di Pisa, Pisa
  - Universita' Campus Bio-medico di Roma, Roma
  - Ospedale Casa Sollievo della Sofferenza - Istituto di Ricovero e Cura a Carattere Scientifico Opera di San Pio da Pietrelcina, San Giovanni Rotondo
  - Fondazione del Piemonte per l'Oncologia - IRCC Candiolo D.O. di Ginecologia Oncologica, Strada Provinciale 142 Km 3.95- Candiolo
  - Azienda Ospedaliero-Universitaria di Parma Dipartimento Clinica Chirurgica e Terapia Chirurgica, Via Gramsci, 14 Parma
  - IRCCS Istituto Nazionale per lo Studio e la Cura dei Tumori, Fondazione Giovanni Pascale Dipartimento di Senologia - Struttura Complessa Oncologia Medica Senologica, Via Mariano Semmola Napoli
  - Azienda Ospedaliero Universitaria Policlinico di Modena Unità Semplice di Senologia, Via Pozzo 71, Modena
  - Azienda Ospedaliero Universitaria di Ferrara c/o Ospedale di Cona Sezione di Clinica Chirurgica, Vial Aldo Moro 8, Cona-Ferrara